CLINICAL TRIAL: NCT01861899
Title: Treatment of Sacroiliac Dysfunction With SI-LOK® Sacroiliac Joint Fixation System
Brief Title: Treatment of Sacroiliac Dysfunction With SI-LOK® Sacroiliac Joint Fixation SI-SI-LOK
Status: Completed | Type: Observational
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RGC12-004_PL_C
Record Dates: First submitted 2013-05-21; First posted 2013-05-24 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Joint Dysfunction
Keywords: Sacro-iliac Joint
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SI-Joint Dysfunction: Device- SI-LOK
  Interventions: Device: SI-LOK

INTERVENTIONS:
Device: SI-LOK — Sacro-iliac joint fusion

SUMMARY:
The objective of this study is to gather clinical data on SI-LOK® for the treatment of sacroiliac joint dysfunction.

The purpose of this prospective study is to evaluate clinical and radiographic outcomes, intra-operative parameters, patient satisfaction and work status following a procedure using SI-LOK® for treatment of sacroiliac joint dysfunction with a minimum of three screws.

DETAILED DESCRIPTION:
Clinical Research Forms will be completed at all pre-op, intra-op and post-op visits by either the surgeon, clinical coordinator or patient.

Forms completed by patients will be checked, initialed and dated by the site coordinator.

Data collected will be presented as mean +/- standard deviation. Statistical significance will be evaluated at the P < 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* A maximum age of 70 years
* Diagnosis of SIJ dysfunction
* Ability to provide Informed Consent for study participation and to return for all follow-up visits

Exclusion Criteria:

* Previous documentation of osteopenia or osteomalacia
* History of metabolic bone disease (e.g. diabetes requiring daily insulin)
* Diagnosis of a condition or requires postoperative medication(s), which may interfere with bony/soft tissue healing
* Presence of a disease entity or condition which totally precludes possibility of bony fusion (e.g. metastatic cancer, HIV, long term use of steroids, etc.)
* History of substance abuse (drugs or alcohol)
* Condition that would preclude completing patient self assessment questionnaires
* Mentally incompetent or prisoner
* Currently a participant in another study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened according to inclusion/exclusion criteria and will be selected for the treatment using the SI-LOK® system
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Radiographic Evaluation | 2 years
  Fusion Assessment Radiolucency

SECONDARY OUTCOMES:
Hospitalization Data | Intra-Operative
  Operative Time Blood Loss Blood Transfusion Hospitalization Time

OTHER OUTCOMES:
Composite of Patient Self-Assessments | 2 years
  Back and Leg Pain Measured by Visual Analog Scale Oswestry Disability Index (ODI) Patient Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Barnum, MD, Principal Investigator — Northwestern Medical Center, St Albans, VT 05478
Locations (1):
- Northwestern Medical Center, Saint Albans, Vermont, United States

IPD SHARING:
Plan to Share IPD: No